CLINICAL TRIAL: NCT05049889
Title: Screening for Individual Susceptibility Factors to Immersion Pulmonary Edema
Acronym: RFSI-OPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2019PBMD07; 2021-A01225-36 (Other: IDRCB)
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The model includes 2 groups:
  * 1 group of divers with a history of immersion pulmonary edema
  * 1 group of matched divers without a history of immersion pulmonary edema
Who Masked: Outcomes Assessor
Masking Description: The investigator who will be in charge of the physiological examination will not know the subject's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- History of Immersion Pulmonary Edema (Active Comparator): The participants will have 2 visits:
  At visit 1 (Day 0), the participants will perform a terrestrial exercise, have a transthoracic cardiac ultrasound, a transthoracic pulmonary ultrasound and several blood samples will be collected.
  At visit 2 (Day 7), the participants will perform a swimming exercise, have a transthoracic cardiac ultrasound, a transthoracic pulmonary ultrasound and several blood samples will be collected.
  Interventions: Other: Terrestrial exercise; Other: Swimming exercise; Device: Transthoracic cardiac ultrasound; Device: Transthoracic pulmonary ultrasound; Biological: Blood collection
- No history of Immersion Pulmonary Edema (Active Comparator): The participants will have 2 visits:
  At visit 1 (Day 0), the participants will perform a terrestrial exercise, have a transthoracic cardiac ultrasound, a transthoracic pulmonary ultrasound and several blood samples will be collected.
  At visit 2 (Day 7), the participants will perform a swimming exercise, have a transthoracic cardiac ultrasound, a transthoracic pulmonary ultrasound and several blood samples will be collected.
  Interventions: Other: Terrestrial exercise; Other: Swimming exercise; Device: Transthoracic cardiac ultrasound; Device: Transthoracic pulmonary ultrasound; Biological: Blood collection

INTERVENTIONS:
Other: Terrestrial exercise — At visit 1 (Day 0), an exercise test will be performed (maximal incremental test), followed by a 30-minute submaximal exercise at constant load.
  During this exercise, continuous data collection will be performed:
  * Continuous 12-lead electrocardiogram
  * Continuous monitoring of blood pressure and ventilation.
Other: Swimming exercise — At visit 2 (Day 7), the subjects will perform a swimming exercise in the experimental pool equipped with a turbine to create a counter-current. The water speed will be constant (4 min per 100 m, i.e. 1.5 km/h). The duration of the exercise will be 30 minutes. Each diver will breathe with the help of a snorkel.
  During this exercise, continuous data collection will be performed:
  * Continuous 12-lead electrocardiogram
  * Continuous monitoring of blood pressure and ventilation.
Device: Transthoracic cardiac ultrasound — The participants will have a transthoracic cardiac ultrasound to measure the dilatations of the cardiac cavities at visit 1 and 2.
Device: Transthoracic pulmonary ultrasound — The participants will have a transthoracic pulmonary ultrasound to quantify the presence of signs of pulmonary vascular overload (comet tails) at visit 1 and 2.
Biological: Blood collection — Several blood samples will be collected at visit 1 and 2.

SUMMARY:
Immersion Pulmonary Edema (IPE) is a relatively new form of hemodynamic pulmonary edema. The number of cases has been increasing over the last ten years and it has become the second most common cause of hospitalization for military divers, after decompression sickness. The pathophysiological mechanisms of IPE are not completely known. Its occurrence is linked to a combination of factors related to the environmental constraints of diving, as well as to the diver's equipment. The main external factors are increased hydrostatic pressure, cold, intense effort and emotional stress. The impact of internal factors is not known. At this time, no severe forms of IPE have been identified in the military. However, it is important to identify this pathology at an early stage, even if the signs appear minor, because the continuation of underwater activity can significantly worsen the clinical picture. The risk of recurrence (greater than 15%) could result in a severe or even lethal accident.

ELIGIBILITY:
Inclusion Criteria:

* Military or civilian diver with at least 100 dives
* Between the ages of 18 and 60
* Good physical condition (able to run/swim for 30 minutes at a constant pace).

Exclusion Criteria:

* Divers with a current temporary medical incapacity to dive
* Persons with contraindications to physical exercise and/or scuba diving
* Pregnant or breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic modifications of the cardiac cavities after exercise | Until the end of the study (49 months)
  The hemodynamic modifications of the cardiac cavities (before/after exercise) will be measured with transthoracic cardiac ultrasound.
Ventilatory regimes | Until the end of the study (49 months)
  Ventilation regimes will be measured with transthoracic pulmonary ultrasound.
Pulmonary compliance | Until the end of the study (49 months)
  Ventilation regimes will be measured with transthoracic pulmonary ultrasound.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Equipe Résidente de Recherche Subaquatique Opérationnelle, Toulon
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided